CLINICAL TRIAL: NCT05322824
Title: Clinical Registration Study of Patients With Intracranial / Carotid Stenosis
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: ROSE
Record Dates: First submitted 2022-04-01; First posted 2022-04-12 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Cognitive Function; Stenosis
Keywords: Cognitive Function; Intracranial / Carotid Stenosis
MeSH Terms: conditions — Constriction, Pathologic; Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: standard medical treatment — standard medical treatment
Procedure: Interventional stenting — Interventional stenting

SUMMARY:
Through prospective registration and follow-up, this study will collect data of patients with intracranial/carotid stenosis, including clinical information, neuropsychological scales, multimodal magnetic resonance images. The investigators aim to analyze clinical and imaging characteristics of patients with cognitive impairment related to intracranial/carotid stenosis, in order to achieve early identification of cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 40 years
* ≥ 50% stenosis in unilateral intracranial / carotid artery
* Written informed consent available

Exclusion Criteria:

* Previous history of major head trauma and any intracranial surgery
* Intracranial abnormalities, such as intracerebral hemorrhage, subarachnoid hemorrhage and other space occupying lesions
* Extrapyramidal symptoms or mental illness which may affect neuropsychological measurement
* Severe loss of vision, hearing, or communicative ability

Exit Criteria:

* Not meet the inclusion criteria
* For any poor adherence, not comply with the requirements of the follow-up, or safety reasons determined by investigator
* Any adverse or serious adverse events during the study period judged by investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intracranial / carotid stenosis aged ≥ 40 years
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the scores of Mini-mental State Examination | 2 years
  Total score of 30. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Incidence of stroke event including ischemic and hemorrhagic stroke | 2 years
Changes in cerebral glymphatic function | 2 years
  assessed by non-invasive diffusion tensor image analysis along the perivascular space (ALPS-index)
Changes in the scores of Montreal Cognitive Assessment | 2 years
  Total score of 30
Changes in cerebral blood flow in the territory of the culprit artery | 2 years
Changes in the scores of Colour Trail Test | 2 years
Changes in the scores of Hopkins Verbal Learning Test | 2 years
Changes in the scores of clock drawing test | 2 years
Changes in the scores of Animal Fluency Test | 2 years
Changes in the scores of Olfactory stick test | 2 years
Changes in metabonomics | 2 years
  include blood and fecal samples

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affilated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China